CLINICAL TRIAL: NCT04393896
Title: Assessing a WeChat-based Integrative Family Intervention (WIFI) for Schizophrenia: a Stepped-wedge Cluster Randomized Trial
Brief Title: Assessing a WeChat-based Integrative Family Intervention (WIFI) for Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 71804197
Record Dates: First submitted 2020-01-27; First posted 2020-05-19 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Family intervention; WeChat; Stepped wedge; Psycho-education; Peer support; Professional support
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster randomized trial. The WeChat-based integrative family intervention (WIFI) program will be implemented in 12 communities affiliated with the Changsha psychiatric hospital through the free medicine delivery process in the 686 Program. The 12 communities will be randomized to one of four fixed sequences every two months during an 8-month intervention period in four clusters of 3 communities each. All clusters will receive the usual financial benefit of the Reward Policy as the control condition, and then successively and in random order, will cross over to the WIFI intervention at 2-month intervals until the study ends.
Who Masked: Outcomes Assessor
Masking Description: people living with schizophrenia, family caregivers, psychiatrists and researchers cannot be blinded for the allocated treatment. The program team conducting the intervention will not be involved in assessing any of the outcomes. The analyses of the data by the researcher will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in the intervention group will receive the usual financial benefits of the Reward Policy as well as the WIFI program which will include three key components: psycho-education through WOA publications, peer-support through a WeChat chat group, and professional support through WeChat private chat and video call.
  Interventions: Behavioral: WeChat-based integrative family intervention (WIFI)
- control group (No Intervention): Participants in the control group will receive the usual financial benefits of the Reward Policy and receive payment from the Changsha psychiatric hospital. However, they will not have access to the WIFI program since they cannot scan the WeChat barcode for the research.

INTERVENTIONS:
Behavioral: WeChat-based integrative family intervention (WIFI) — The WIFI program will include three key components: psycho-education through WeChat Official Account publications, peer-support through a WeChat chat group, and professional support through WeChat private chat and video call
  Arms: intervention group

SUMMARY:
The study aims to test both the effectiveness and implementation strategy of a WeChat-based integrative family intervention (WIFI) to support family caregiving of schizophrenia in China.

DETAILED DESCRIPTION:
The investigators will conduct a type 2 hybrid effectiveness-implementation study to test both the effect of and the implementation process of a WeChat-based integrative family intervention (WIFI) program. The program will include three core components: 1) psycho-education through WeChat Official Account (WOA), 2) peer support through WeChat chat group, and 3) professional support through WeChat video chat. A rigorous stepped wedge cluster randomized trial will be used to evaluate the implementation, effectiveness, and cost of the WIFI program. The WIFI program will be implemented in 12 communities affiliated with the Changsha psychiatric hospital through the free medicine delivery process in the 686 Program. 20 families of schizophrenia will be selected from each community. The 12 communities will be randomized to one of four fixed sequences every two months during an 8-month intervention period in four clusters of 3 communities each. All clusters will receive the usual financial benefit of the Reward Policy as the control condition, and then successively and in random order, will cross over to the WIFI program at 2-month intervals until the study ends. Outcomes will be assessed for both family caregivers and the family member with schizophrenia. Family caregivers will be assessed for their knowledge and skills about caregiving, social support and coping, perceived stigma, caregiver burden, family functioning, positive feelings, and psychological distress. Schizophrenia individuals will be assessed for their symptoms and functioning, quality of life, recovery and re-hospitalization. Cost data such as costs of the intervention, health care utilization, and costs associated with lost productivity will also be collected. In addition, the investigators will collect process data including fidelity and quality of program implementation as well as users' attitudes will also be collected. Treatment effects will be estimated using generalized linear maximum likelihood mixed modeling (GLMM) with clusters as a random effect and time as a fixed effect. Cost-effectiveness analysis will be performed from the societal perspective using incremental cost effectiveness ratios (ICERs). Qualitative analysis will use the grounded theory approach and immersion-crystallization process. All statistical analyses will be conducted according to the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

For people living with schizophrenia:

* being registered in the "686 Program"
* fulfilling the Chinese Classification of Mental Disorders-3 (CCMD-3) or the International Classification of Diseases-10 (ICD-10) criteria for schizophrenia
* living with at least one family member
* able to use a smartphone and WeChat to read and communicate

For family members:

* joining the Reward Policy and receiving a subsidy for family care
* living with schizophrenia individuals for at least the past two years
* involved with caregiving activities of schizophrenia individuals
* able to use a smartphone and WeChat to read and communicate
* at least one family member having a smartphone with WeChat app installed.

Exclusion Criteria:

For people living with schizophrenia:

* diagnosed with mental illness other than schizophrenia
* living alone with no family members
* not able to use smartphones or WeChat

For family members:

* not involved with caregiving activities for the schizophrenia individuals
* not able to use smartphones or WeChat

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
caregiver burden at baseline | baseline
  caregiver burden will be measured using the internationally standard caregiving burden scale---Zarit Burden Interview (ZBI) at baseline. The total score ranges from 0 to 88, with higher composite score indicating higher caregiver burden.
caregiver burden at month 2 | 2 months
  caregiver burden will be measured using the internationally standard caregiving burden scale---Zarit Burden Interview (ZBI) after 2 months. The total score ranges from 0 to 88, with higher composite score indicating higher caregiver burden.
caregiver burden at month 4 | 4 months
  caregiver burden will be measured using the internationally standard caregiving burden scale---Zarit Burden Interview (ZBI) after 4 months. The total score ranges from 0 to 88, with higher composite score indicating higher caregiver burden.
caregiver burden at month 6 | 6 months
  caregiver burden will be measured using the internationally standard caregiving burden scale---Zarit Burden Interview (ZBI) after 6 months. The total score ranges from 0 to 88, with higher composite score indicating higher caregiver burden.
caregiver burden at month 8 | 8 months
  caregiver burden will be measured using the internationally standard caregiving burden scale---Zarit Burden Interview (ZBI) after 8 months. The total score ranges from 0 to 88, with higher composite score indicating higher caregiver burden.

SECONDARY OUTCOMES:
Depression | 8 months
  Depression will be measured using the internationally standard depression scale---Patient Health Questionnaire-9 (PHQ-9) at baseline, 2 months, 4 months, 6 months, 8 months. The total score ranges from 0 to 27, with higher score indicating more depressive symptoms.
Anxiety | 8 months
  Anxiety will be measured using the internationally standard anxiety scale---Generalized Anxiety Disorder Scale-7 (GAD-7) at baseline, 2 months, 4 months, 6 months, 8 months. The total score ranges from 0 to 27, with higher score indicating more anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Yu, PhD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the official start of the trial to the end of the trial
Access Criteria: Describe clearly about the reason of review

REFERENCES:
- [Background] Yu Y, Liu ZW, Tang BW, Zhao M, Liu XG, Xiao SY. Reported family burden of schizophrenia patients in rural China. PLoS One. 2017 Jun 19;12(6):e0179425. doi: 10.1371/journal.pone.0179425. eCollection 2017. PMID 28628657
- [Background] Yu Y, Liu ZW, Zhou W, Chen XC, Zhang XY, Hu M, Xiao SY. Assessment of Burden Among Family Caregivers of Schizophrenia: Psychometric Testing for Short-Form Zarit Burden Interviews. Front Psychol. 2018 Dec 19;9:2539. doi: 10.3389/fpsyg.2018.02539. eCollection 2018. PMID 30618960
- [Background] Yu Y, Tang BW, Liu ZW, Chen YM, Zhang XY, Xiao S. Who cares for the schizophrenia individuals in rural China - A profile of primary family caregivers. Compr Psychiatry. 2018 Jul;84:47-53. doi: 10.1016/j.comppsych.2018.04.002. Epub 2018 Apr 11. PMID 29684660
- [Background] Yu Y, Zhou W, Xiao S. China's Reward Policy for Family Care of Persons With Serious Mental Illness. Psychiatr Serv. 2018 Dec 1;69(12):1210-1211. doi: 10.1176/appi.ps.201800114. Epub 2018 Oct 18. PMID 30332924
- [Background] Yu Y, Zhou W, Liu ZW, Hu M, Tan ZH, Xiao SY. Gender differences in caregiving among a schizophrenia population. Psychol Res Behav Manag. 2018 Dec 20;12:7-13. doi: 10.2147/PRBM.S187975. eCollection 2019. PMID 30588138
- [Derived] Yu Y, Li T, Xi S, Li Y, Xiao X, Yang M, Ge X, Xiao S, Tebes J. Assessing a WeChat-Based Integrative Family Intervention (WIFI) for Schizophrenia: Protocol for a Stepped-Wedge Cluster Randomized Trial. JMIR Res Protoc. 2020 Aug 25;9(8):e18538. doi: 10.2196/18538. PMID 32687478